CLINICAL TRIAL: NCT06195163
Title: Transdermal Testosterone Pretreatment in Poor Responders With Androgen Receptor Polymorphism Undergoing ICSI: A Randomized Clinical Investigation.
Brief Title: TRAP Study: Testosterone for Androgen Receptor Polymorphism
Acronym: TRAP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Bernabeu (Other)
Responsible Party: Principal Investigator, Andrea Bernabeu García, Principal Investigator, Instituto Bernabeu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBMR46
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Fertility Disorders
Keywords: ovarian stimulation; testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental): Daily 10 mg transdermal testosterone for 21 days prior to the start of ovarian stimulation.
  Interventions: Drug: Transdermal Gel in Sachet Dosage Form
- Control group (Active Comparator): No pre-treatment prior to ovarian stimulation.
  Interventions: Drug: No pretreatment

INTERVENTIONS:
Drug: Transdermal Gel in Sachet Dosage Form — Transdermal testosterone gel application prior to ovarian stimulation in the study group.
  Arms: Study group
Drug: No pretreatment — No pretreatment prior to the ovarian stimulation in the control group.
  Arms: Control group

SUMMARY:
To determine whether pretreatment with transdermal testosterone increases the number of cumulus-oocyte complexes (COCs) obtained after ovarian stimulation by more than 1.5 in patients with low ovarian reserve and androgen receptor polymorphism undergoing intracytoplasmic sperm injection (ICSI).

ELIGIBILITY:
Inclusion Criteria:

* Patients with low ovarian reserve according to Bologna criteria: at least two of the following three:

  1. Age equal to or greater than 40 years.
  2. Previous cycle with less than 4 oocytes retrieved.
  3. Low ovarian reserve markers (antral follicle count <5-7; AMH <0.5-1.1 ng).
* Carriers of androgen receptor polymorphism: between 22 and 24 CAG repeats.
* Body Mass Index (BMI) less than 32.
* Indication for in vitro fertilization.
* Presence of both ovaries.
* Absence of ovarian cysts.
* Absence of endometriosis.
* Normal karyotype and fragile X study.
* Absence of severe male factor.
* Semen sample from ejaculate.
* Ability to comply with the study protocol.
* To have given written consent.

Exclusion Criteria:

* Non-compliance with instructions or non-formalization of informed consent.
* Concurrent participation in another study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of COC (cumulus-oocyte complexes) | Egg collection day (between 8 and 14 days after starting of ovarian stimulation)
  If number of COC is higher at least by 1.5 in the experimental group.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Bernabeu, Alicante, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barbieri RL, Sluss PM, Powers RD, McShane PM, Vitonis A, Ginsburg E, Cramer DC. Association of body mass index, age, and cigarette smoking with serum testosterone levels in cycling women undergoing in vitro fertilization. Fertil Steril. 2005 Feb;83(2):302-8. doi: 10.1016/j.fertnstert.2004.07.956. PMID 15705366
- [Background] Bosdou JK, Venetis CA, Dafopoulos K, Zepiridis L, Chatzimeletiou K, Anifandis G, Mitsoli A, Makedos A, Messinis IE, Tarlatzis BC, Kolibianakis EM. Transdermal testosterone pretreatment in poor responders undergoing ICSI: a randomized clinical trial. Hum Reprod. 2016 May;31(5):977-85. doi: 10.1093/humrep/dew028. Epub 2016 Mar 7. PMID 26956551
- [Background] Bosdou JK, Venetis CA, Kolibianakis EM, Toulis KA, Goulis DG, Zepiridis L, Tarlatzis BC. The use of androgens or androgen-modulating agents in poor responders undergoing in vitro fertilization: a systematic review and meta-analysis. Hum Reprod Update. 2012 Mar-Apr;18(2):127-45. doi: 10.1093/humupd/dmr051. Epub 2012 Feb 3. PMID 22307331
- [Background] Drakopoulos P, Bardhi E, Boudry L, Vaiarelli A, Makrigiannakis A, Esteves SC, Tournaye H, Blockeel C. Update on the management of poor ovarian response in IVF: the shift from Bologna criteria to the Poseidon concept. Ther Adv Reprod Health. 2020 Jul 31;14:2633494120941480. doi: 10.1177/2633494120941480. eCollection 2020 Jan-Dec. PMID 32844159
- [Background] Duffy JMN, Bhattacharya S, Bhattacharya S, Bofill M, Collura B, Curtis C, Evers JLH, Giudice LC, Farquharson RG, Franik S, Hickey M, Hull ML, Jordan V, Khalaf Y, Legro RS, Lensen S, Mavrelos D, Mol BW, Niederberger C, Ng EHY, Puscasiu L, Repping S, Sarris I, Showell M, Strandell A, Vail A, van Wely M, Vercoe M, Vuong NL, Wang AY, Wang R, Wilkinson J, Youssef MA, Farquhar CM; Core Outcome Measure for Infertility Trials (COMMIT) initiative. Standardizing definitions and reporting guidelines for the infertility core outcome set: an international consensus development study. Fertil Steril. 2021 Jan;115(1):201-212. doi: 10.1016/j.fertnstert.2020.11.013. Epub 2020 Nov 30. PMID 33272619
- [Background] Ferraretti AP, La Marca A, Fauser BC, Tarlatzis B, Nargund G, Gianaroli L; ESHRE working group on Poor Ovarian Response Definition. ESHRE consensus on the definition of 'poor response' to ovarian stimulation for in vitro fertilization: the Bologna criteria. Hum Reprod. 2011 Jul;26(7):1616-24. doi: 10.1093/humrep/der092. Epub 2011 Apr 19. PMID 21505041
- [Background] Laisk T, Haller-Kikkatalo K, Laanpere M, Jakovlev U, Peters M, Karro H, Salumets A. Androgen receptor epigenetic variations influence early follicular phase gonadotropin levels. Acta Obstet Gynecol Scand. 2010 Dec;89(12):1557-63. doi: 10.3109/00016349.2010.526182. Epub 2010 Nov 5. PMID 21050150
- [Background] Lledo B, Llacer J, Ortiz JA, Martinez B, Morales R, Bernabeu R. A pharmacogenetic approach to improve low ovarian response: The role of CAG repeats length in the androgen receptor gene. Eur J Obstet Gynecol Reprod Biol. 2018 Aug;227:41-45. doi: 10.1016/j.ejogrb.2018.06.001. Epub 2018 Jun 4. PMID 29886316
- [Background] Lledo B, Llacer J, Turienzo A, Ortiz JA, Guerrero J, Morales R, Ten J, Bernabeu R. Androgen receptor CAG repeat length is associated with ovarian reserve but not with ovarian response. Reprod Biomed Online. 2014 Oct;29(4):509-15. doi: 10.1016/j.rbmo.2014.06.012. Epub 2014 Jul 9. PMID 25131556
- [Background] Lledo B, Ortiz JA, Llacer J, Bernabeu R. Pharmacogenetics of ovarian response. Pharmacogenomics. 2014 Apr;15(6):885-93. doi: 10.2217/pgs.14.49. PMID 24897293
- [Background] Subira J, Algaba A, Vazquez S, Taroncher Dasi R, Molla Robles G, Monzo Fabuel S, Baydal V, Ruiz Herreros A, Garcia Camunas N, Rubio Rubio JM. Testosterone does not improve ovarian response in Bologna poor responders: a randomized controlled trial (TESTOPRIM). Reprod Biomed Online. 2021 Sep;43(3):466-474. doi: 10.1016/j.rbmo.2021.05.021. Epub 2021 May 30. PMID 34312088
- [Background] Sunkara SK, Rittenberg V, Raine-Fenning N, Bhattacharya S, Zamora J, Coomarasamy A. Association between the number of eggs and live birth in IVF treatment: an analysis of 400 135 treatment cycles. Hum Reprod. 2011 Jul;26(7):1768-74. doi: 10.1093/humrep/der106. Epub 2011 May 10. PMID 21558332
- [Background] Vendola KA, Zhou J, Adesanya OO, Weil SJ, Bondy CA. Androgens stimulate early stages of follicular growth in the primate ovary. J Clin Invest. 1998 Jun 15;101(12):2622-9. doi: 10.1172/JCI2081. PMID 9637695